CLINICAL TRIAL: NCT04849520
Title: Effect of High-flow Nasal Oxygenation on Safe Apnea Time in Children With Open Mouth
Brief Title: High Flow Nasal Cannula for Safe Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Principal Investigator, Jin-Tae Kim, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2102-149-1200
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia, General; Apnea
Keywords: Oxygenation; High-flow nasal cannula
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High flow (Experimental): Application of high flow nasal cannula during apnea
  Interventions: Device: High flow nasal cannula
- Buccal (Active Comparator): Application of buccal oxygenation during apnea
  Interventions: Device: Buccal oxygenation

INTERVENTIONS:
Device: High flow nasal cannula — Oxygen supplement via high flow nasal cannula at a rate of 2 liters/kg/min
  Arms: High flow
Device: Buccal oxygenation — Oxygen supplement intra-orally via oral Ring-Adair-Elwyn endotracheal tube connected to oxygen at a rate of 0.5 liters/kg/min
  Arms: Buccal

SUMMARY:
This is a prospective randomized controlled trial comparing high flow nasal cannula and buccal oxygenation as method of oxygenation during apnea in children.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial comparing two oxygenation methods for prolongation of apnea time in children aged 0 to 10 years old.

This study measures time for the pulse oximetry drop from 100% to 92% after oxygenation with 100% oxygen, applying high flow nasal cannula or buccal oxygen insufflation via an oral Ring-Adair-Elwyn endotracheal tube connected to oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Children under 11 years old undergoing general anesthesia with American Society of Anesthesiologists Physical Status 1 or 2.

Exclusion Criteria:

* Refusal of enrollment from one or more legal guardians of the patient
* Plan of usage of supraglottic airway device as airway maintenance device
* Presence of upper respiratory tract infection of lung disease
* Premature infants younger than postconceptual age of 40 weeks
* Anticipation of difficult bag-mask ventilation due to facial anomaly or micrognathia
* Other conditions that are considered inappropriate for the study

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Apnea success rate | From start of apnea to drop of pulse oximetry to 92%, up to 520 seconds
  Proportion of patients that succeed in prolongation of apnea time while maintaining pulse oximetry > 92%

SECONDARY OUTCOMES:
Apnea time | From start of apnea to drop of pulse oximetry to 92%, up to 520 seconds
  Time elapsed from start of apnea to resume of bag-mask ventilation
End-tidal carbon dioxide | After resuming of bag-mask ventilation, up to 30 seconds
  End-tidal carbon dioxide partial pressure of first resumed breath after apnea
Minimal pulse oximetry | After resuming of bag-mask ventilation, up to 60 seconds
  Lowest value of pulse oximetry after resume of bag-mask ventilation
Time to pulse oximetry of 100 percent | After resuming of bag-mask ventilation, up to 300 seconds
  Time elapsed from resume of bag-mask ventilation to regain of 100 percent in the pulse oximetry value
Electrocardiogram | From start of study to end of study, up to 20 min
  Appearance of any arrhythmia or prolonged QT interval measured throughout the study
Mean blood pressure | From start of study to end of study, up to 20 min
  Mean non-invasive blood pressure measured throughout the study
Pulse oximetry | From start of study to end of study, up to 20 min
  Pulse oximetry measured throughout the study
Oxygen reserve index | From start of study to end of study, up to 20 min
  Oxygen reserve index measured throughout the study
Transcutaneous carbon dioxide | From start of study to end of study, up to 20 min
  Transcutaneous carbon dioxide level measured throughout the study
Heart rate | From start of study to end of study, up to 20 min
  Heart rate measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Frei FJ, Ummenhofer W. Difficult intubation in paediatrics. Paediatr Anaesth. 1996;6(4):251-63. doi: 10.1111/j.1460-9592.1996.tb00447.x. No abstract available. PMID 8827740
- [Background] Schibler A, Hall GL, Businger F, Reinmann B, Wildhaber JH, Cernelc M, Frey U. Measurement of lung volume and ventilation distribution with an ultrasonic flow meter in healthy infants. Eur Respir J. 2002 Oct;20(4):912-8. doi: 10.1183/09031936.02.00226002. PMID 12412683
- [Background] King W, Petrillo T, Pettignano R. Enteral nutrition and cardiovascular medications in the pediatric intensive care unit. JPEN J Parenter Enteral Nutr. 2004 Sep-Oct;28(5):334-8. doi: 10.1177/0148607104028005334. PMID 15449573
- [Background] Schibler A, Yuill M, Parsley C, Pham T, Gilshenan K, Dakin C. Regional ventilation distribution in non-sedated spontaneously breathing newborns and adults is not different. Pediatr Pulmonol. 2009 Sep;44(9):851-8. doi: 10.1002/ppul.21000. PMID 19672959
- [Background] Schibler A, Henning R. Positive end-expiratory pressure and ventilation inhomogeneity in mechanically ventilated children. Pediatr Crit Care Med. 2002 Apr;3(2):124-128. doi: 10.1097/00130478-200204000-00006. PMID 12780980
- [Background] Erb T, Marsch SC, Hampl KF, Frei FJ. Teaching the use of fiberoptic intubation for children older than two years of age. Anesth Analg. 1997 Nov;85(5):1037-41. doi: 10.1097/00000539-199711000-00013. PMID 9356095
- [Background] Mir F, Patel A, Iqbal R, Cecconi M, Nouraei SA. A randomised controlled trial comparing transnasal humidified rapid insufflation ventilatory exchange (THRIVE) pre-oxygenation with facemask pre-oxygenation in patients undergoing rapid sequence induction of anaesthesia. Anaesthesia. 2017 Apr;72(4):439-443. doi: 10.1111/anae.13799. Epub 2016 Dec 30. PMID 28035669
- [Background] Lodenius A, Piehl J, Ostlund A, Ullman J, Jonsson Fagerlund M. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) vs. facemask breathing pre-oxygenation for rapid sequence induction in adults: a prospective randomised non-blinded clinical trial. Anaesthesia. 2018 May;73(5):564-571. doi: 10.1111/anae.14215. Epub 2018 Jan 13. PMID 29330853
- [Background] Humphreys S, Lee-Archer P, Reyne G, Long D, Williams T, Schibler A. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) in children: a randomized controlled trial. Br J Anaesth. 2017 Feb;118(2):232-238. doi: 10.1093/bja/aew401. PMID 28100527
- [Background] Lyons C, Callaghan M. Uses and mechanisms of apnoeic oxygenation: a narrative review. Anaesthesia. 2019 Apr;74(4):497-507. doi: 10.1111/anae.14565. Epub 2019 Feb 19. PMID 30784037
- [Background] Wettstein RB, Shelledy DC, Peters JI. Delivered oxygen concentrations using low-flow and high-flow nasal cannulas. Respir Care. 2005 May;50(5):604-9. PMID 15871753
- [Background] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404
- [Background] Heard A, Toner AJ, Evans JR, Aranda Palacios AM, Lauer S. Apneic Oxygenation During Prolonged Laryngoscopy in Obese Patients: A Randomized, Controlled Trial of Buccal RAE Tube Oxygen Administration. Anesth Analg. 2017 Apr;124(4):1162-1167. doi: 10.1213/ANE.0000000000001564. PMID 27655276